CLINICAL TRIAL: NCT00088530
Title: Pixantrone (BBR 2778) Versus Other Chemotherapeutic Agents for Third-line Single Agent Treatment of Patients With Relapsed Aggressive Non-Hodgkin's Lymphoma: A Randomized, Controlled, Phase III Comparative Trial
Brief Title: BBR 2778 for Relapsed, Aggressive Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIX301; NCT00101049 (obsolete NCT alias)
Record Dates: First submitted 2004-07-28; First posted 2004-07-29 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Pixantrone; Non-Hodgkins lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pixantrone; Cyclophosphamide; Vincristine; Rituximab; Prednisone; Vinorelbine; Etoposide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm (Experimental): Pixantrone (BBR2778)
  Interventions: Drug: pixantrone, cyclophosphamide, vincristine, rituximab, prednisone
- Comparator Arm (Active Comparator): To be chosen by the investigator, among vinorelbine, oxaliplatin, ifosfamide, etoposide or mitoxantrone
  Interventions: Drug: Vinorelbine, Oxalplatin, Ifosfasmide, Etoposide, Mitoxatrone, Gemcitabine or Rituximab

INTERVENTIONS:
Drug: pixantrone, cyclophosphamide, vincristine, rituximab, prednisone — Day 1: pixantrone (150 mg/m2), cyclophosphamide (750 mg/m2), vincristine (1.4 mg/m2), rituximab (375 mg/m2) Days 1-5: prednisone (100 mg/day)
  Other Names: BBR2778
  Arms: Experimental Arm
Drug: Vinorelbine, Oxalplatin, Ifosfasmide, Etoposide, Mitoxatrone, Gemcitabine or Rituximab — Day 1: cyclophosphamide (750 mg/m2), vincristine (1.4 mg/m2), rituximab (375 mg/m2) Days 1-5: prednisone (100 mg/day)
  Arms: Comparator Arm

SUMMARY:
BBR 2778 is a novel aza-anthracenedione that has activity in experimental tumors and shows reduced potential for cardiotoxicity in animal models. This cytotoxic agent has structural similarities with mitoxantrone as well as general similarities with anthracyclines (such as the tricyclic central quinoid chromophore).

DETAILED DESCRIPTION:
The primary study objective is to compare the efficacy of BBR 2778 to a selection of single agents. Secondary objectives are to compare the safety and tolerability of BBR 2778 to a selection of single agents, and to assess the pharmacokinetic parameters of BBR 2778 in a subset of this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aggressive [de novo or transformed] NHL according to REAL/WHO classification.
* At least one objectively measurable lesion as demonstrated by CT, spiral CT, or MRI and plain radiograph of the chest (chest x-ray, for chest lesions only) that can be followed for response as target lesion.
* Relapse after 2 or more prior regimens of chemotherapy
* ECOG performance status of 0, 1, or 2
* Adequate hematologic, renal and hepatic function
* LVEF ≥50% determined by MUGA scan

Exclusion Criteria:

* Prior treatment with a cumulative dose of doxorubicin or equivalent exceeding 450 mg/m²
* Prior allogenic stem cell transplant
* Histological diagnosis of Burkitt lymphoma, lymphoblastic lymphoma or Mantle cell lymphoma
* Active CNS lymphoma or HIV-related lymphoma.
* Any chemotherapy, radiotherapy, or other anticancer treatment (including corticosteroid, 10 or more mg/day of prednisone or equivalent) within the 2 weeks before randomization
* Pregnant women or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-07; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simran Singh, Study Director — Sr. Director, Clinical Operations
Locations (99):
- United States (9):
  - Robert A. Moss, M.D., FACP, Inc., Fountain Valley, California
  - UCLA Medical Center, Los Angeles, California
  - Watson Clinic for Cancer Care and Research, Lakeland, Florida
  - Rush University Medical Center, Chicago, Illinois
  - New Mexico Oncology/Hematology, Albuquerque, New Mexico
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Northwest Kaiser Permanente, Portland, Oregon
  - Northern Utah Hematology Oncology, P.C., Ogden, Utah
- Argentina (8):
  - Clinica Modelo S.A., Paraná, Entre Ríos Province
  - Instituto de Investigaciones Clinicas, Rosario, Santa Fe Province
  - Centro Oncologico Rosario, Rosario, Santa Fe Province
  - FUNDALEU - fundacion para combatir le Leucernia, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Academia Nacional de Medicina, Caba
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
  - ISIS Clinica Especializada, Santa Fe
- Bulgaria (3):
  - University Gernal Hospital for Active Treatment "Alexandrovska" - Clinic of Hematology, Sofia
  - National Centre for Hemotransfusion, Sofia
  - University General Hospital for Active Treatment "St. Marina" Clinic of Hematology, Varna
- Hospital CIMA San Jose, Escazú, Costa Rica
- Ecuador (3):
  - Hospital Oncologico de Solca, Capilla Mauta, Guayaquil
  - Hospital Carlos Andrade Marin Oncologia, Quito, Pinchincha
  - Hospital Solca Quito, Quito
- Tartu University Clinics, Hematology Oncology Clinic, Tartu, Estonia
- France (3):
  - Institute Bergonie, Bordeaux
  - Centre Hospitalier Lyo Sud, Service d'Hematologie et d'Oncologie, Pierre-Bénite
  - Hopitaux Universitaires de Strabourg - Hopital de Hautepierre, Strasbourg
- Germany (7):
  - Staedtische Kliniken Hoechst, Frankfurt am Main, Hesse
  - Charite, Campus Benjamin Franklin, Berlin
  - Klinikum der Universitaet zu Koeln, Cologne
  - Universitatklinik des Saarlandes, Innere Medzin I, Hamburg
  - Westpfalzklinikum Kaiserslautern, Kaiserslautern
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Mutterhaus der Borromaeerinne, Trier
- Hungary (6):
  - Szent Laszlo Korhaz, Budapest
  - Petz Aladar Megyei Okato Korhaz, Győr
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Kaposi Mor Megyei Korhaz, Kaposvár
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Orvos-es Gyogy II, Szeged
- India (8):
  - Indo-American Cancer Institute & Research Center, Hyderabaad, AndhPrad
  - Nizam's Institute of Medical Sciences, Panjagutta, Hyderabad
  - Manipal Hospital, Bangalore, Karnataka
  - Shirdi Sai Baba Cancer Hospital, K.M.C. Manipal, Manipal, Karna
  - Regional Cancer Center, Thiruvananthapuram, Kerla
  - Bhagwan Mahaveer Cancer Hospital & Research Center, Jaipur, Rajasthan
  - M.S. Ramaiah Medical College, Bangalore
  - Tata Memorial Hospital, Mumbai
- Italy (13):
  - Policlinico S. Orsola, Instituto di Ematologia, Bologna
  - Ospedale Oncologico "A. Businco", Cagliari
  - Ospedale S. Martino, Genova
  - Universita degli Studi Perugia Policlinico Monteluce, Perugia
  - Azienda ospedaliera Pisana "Santa Chiara", Pisa
  - Azienda Ospedaliera Pisanan "Santana Chiara", Pisa
  - Ospedale Oncolgoico Regionale della Basilicata, Rionero in Vulture
  - Ospedale S. Eugenio, Roma
  - Universita La Sapienza, Roma
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Policlinico S. Maria alle Scotte, Siena
  - Presidio San Giuseppe Moscati, Taranto
  - Ospedale Civile, Udine
- Mexico (2):
  - Fundacion Centro De Investigacion, Medellín, Columbia
  - Medical Solutions, Guatemala, Guatemala
- Complejo Hospitalario "Arnulfo Arias Madrid, Panama City, Panama
- Peru (2):
  - Hospital Edgardo Rebagliati Martins, Lima
  - Onococenter, San Borja
- Klinika Hematologii, Onkologii i Chorob Wewnetrznych, Gdansk, Poland
- Romania (6):
  - Brasov Counthy Hospital, Brasov
  - Colentina Clinical Hospital Hem Dept, Bucharest
  - Fundei Clinical Institute, Bucharest
  - Institutul Oncologic "Ion Chiricuta" Oncologie Medicala, Cluj-Napoca
  - Prof. Dr. Ian Chiricuta, Institute of Oncology, Radiotheraphy, Cluj-Napoca
  - Mures County Clinical Hospital, Târgu Mureş
- Russia (16):
  - State Medical Institution Altai Territorial Oncological Center, Barnaul
  - State Medical Institution Replubican Oncological Center, Bashkortostan
  - State Therapeutical & Prophlatic Institution: Cheylabinsk Regional Oncological Center, Chelyabinsk
  - State Medical Institution, Irkutsk
  - State Medical Institution: Clinical Oncological Center, Krasnodar
  - Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - State Institution: Hematological Research Center under the Russian Academy of Medical Sciences, Moscow
  - State Institution: Moscow Regional Research Clinical institute n.a. M.F., Moscow
  - Semashko Central Clinical Hospital, Moscow
  - Medical Radiological Research Center under the Russian academey of Medical Sciences, Obninsk
  - Research Insitute of Hematology and Blood Transfusion, Saint Petersburg
  - St. Petersburg Pavlov State Medical Clinic of Intensive Care & Bone Marrow Transplantation, Saint Petersburg
  - St. Petersburg State Medical univ. n.a. I.P. Pavlov, Saint Petersburg
  - St. Petersburg State Medical Institution: Municipal Hospital #31, Saint Petersburg
  - Central Research Rontgenological and Radiological Institute, Saint Petersburg
  - State Research Institution: Research Institute of Oncology, Saint Petersburg
- Ukraine (4):
  - Institute of Clinical Radiology of the Research Center for Radiation Medicine under the UAMS, Kyiv
  - Kyiv Bone Marrow Transplantation, Kyiv
  - Institute of Blood Pathology & Transfusion Medicine under the UAMS, Lviv
  - Zhtomyr O.F. Gerbachevsky Regional Hospital, Zhytomyr
- United Kingdom (3):
  - Beatson Oncology Centre, Western Infirmary, Glasgow
  - St. Georges Hospital, London
  - Weston Park Hospital, Sheffield
- Uruguay (2):
  - Hospital Maciel, Montevideo
  - Hospital Policial de Montevideo, Poblado Montevideo Chico

REFERENCES:
- [Derived] Pettengell R, Coiffier B, Narayanan G, de Mendoza FH, Digumarti R, Gomez H, Zinzani PL, Schiller G, Rizzieri D, Boland G, Cernohous P, Wang L, Kuepfer C, Gorbatchevsky I, Singer JW. Pixantrone dimaleate versus other chemotherapeutic agents as a single-agent salvage treatment in patients with relapsed or refractory aggressive non-Hodgkin lymphoma: a phase 3, multicentre, open-label, randomised trial. Lancet Oncol. 2012 Jul;13(7):696-706. doi: 10.1016/S1470-2045(12)70212-7. Epub 2012 May 30. PMID 22652183
- See also: CTI company website — http://www.celltherapeutics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 66 sites: 6 in the U.S, 4 in France, 3 in Bulgaria, 4 sites in Hungary, 3 in Ukraine, 11 in Italy, 2 in Romania, 3 in United Kingdom, 2 in Poland, 2 in Germany, 3 in Peru, 6 in Argentina, 1 in Colombia, 2 in Ecuador, 1 in Uruguay, 5 in Russia and 8 in India.
Groups:
- Experimental Group: Pixantrone (BBR 2778) 85 mg/m2 on days 1, 8 and 15 of each 28-day cycle)
- Comparator Group: Vinorelbine or Oxalplatin or Ifosfasmide or Etoposide or Mitoxatrone or Gemcitabine or Rituximab
Period: Overall Study
Arm/Group | Experimental Group | Comparator Group
Started | 70 | 70
Completed | 20 | 16
Not Completed | 50 | 54
Not completed — Progressive/Relapsed Disease | 28 | 39
Not completed — Adverse Event | 15 | 9
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor decision | 0 | 1
Not completed — Patient never treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: Pixantrone (BBR 2778) 85 mg/m2 on days 1, 8 and 15 of each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Comparator Group | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at Randomization (years) | 58.2 (13.5) | 56.2 (12.9) | 57.2 (13.2)
Age, Customized [Count of Participants; unit: Participants]
  18 to < 30 | 5 | 2 | 7
  30 to < 40 | 2 | 9 | 11
  40 to < 50 | 9 | 7 | 16
  50 to < 60 | 18 | 21 | 39
  60 to < 70 | 20 | 21 | 41
  70 to < 80 | 15 | 9 | 24
  ≥ 80 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 46 | 40 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 46 | 44 | 90
  Black | 0 | 0 | 0
  Asian | 10 | 13 | 23
  Hispanic | 7 | 6 | 13
  Native American | 1 | 1 | 2
  Other | 6 | 6 | 12
Region of Enrollment [Number; unit: participants] — Demographic data will be displayed and summary statistics will be used to describe the study population (i.e., means, medians, and ranges of age, weight, and height, and frequencies for race, gender, baseline performance status, and tumor types and histology). No formal statistical tests will be done.
  participants
    North America | 4 | 4 | 8
    Argentina | 6 | 5 | 11
    Bulgaria | 6 | 3 | 9
    Colombia | 1 | 0 | 1
    Ecuador | 3 | 4 | 7
    Hungary | 5 | 5 | 10
    India | 9 | 12 | 21
    Peru | 9 | 8 | 17
    Poland | 2 | 0 | 2
    Romania | 1 | 1 | 2
    Russian Federation | 4 | 5 | 9
    Ukraine | 1 | 3 | 4
    Uruguay | 0 | 1 | 1
    France | 4 | 4 | 8
    United Kingdom | 4 | 3 | 7
    Germany | 3 | 0 | 3
    Italy | 8 | 12 | 20
Baseline ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Grade as published in Oken MM, et al. ECOG PS grade 0- Fully active, able to carry on all predisease performance without restriction; 1 - restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; 2- ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3- capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  Participants
    0 | 26 | 23 | 49
    1 | 30 | 32 | 62
    2 | 14 | 14 | 28
    3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) and Complete Response Unconfirmed (CRu)
Description: Proportion of patients with a best response of complete response (CR) or Complete Response unconfirmed (CRu) in the End Of Treatment (EOT) or End Of Study (EOS) analyses by independent assessment in the Intent-to-treat (ITT) population through the End of Treatment (EOT)
Time Frame: EOT; approximately 6 months
Population: Intent to Treat (all randomized patients)
Measure: Number (95% Confidence Interval); unit: percentage of randomized patients
Arm/Group | Experimental Group | Comparator Group
Number analyzed (Participants) | 70 | 70
percentage of randomized patients
  END OF TREATMENT: CR/CRu, n (%) | 20.0 [11.4 to 31.3] | 5.7 [1.6 to 14.0]
  END OF STUDY: CR/CRu, n (%) | 24.3 [14.8 to 36.0] | 7.1 [2.4 to 15.9]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The time between the date of randomization and the date of the initial documentation of progressive/relapsed disease or death due to any cause.
Time Frame: 18 months after 6 cycles of treatment; approximately 24 months
Population: Intent-to-treat patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Group | Comparator Group
Number analyzed (Participants) | 70 | 70
months | 5.3 [2.3 to 6.2] | 2.6 [1.9 to 3.5]

3. Secondary Outcome: Overall Survival
Description: The time between the date of randomization and the date of death due to any cause.
Time Frame: 18 months after 6 cycles of treatment; approximately 24 months
Population: Intent-To-Treat (ITT) Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Group | Comparator Group
Number analyzed (Participants) | 70 | 70
Months | 10.2 [6.4 to 15.7] | 7.6 [5.4 to 9.3]

4. Secondary Outcome: Overall Response Rate (ORR) Lasting at Least 4 Months
Description: The proportion of patients with Complete response or Partial Response with a difference from the first documented objective response to disease progression or death of at least 4 months.
Time Frame: approximately 24 months
Population: Intent-To-Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Experimental Group | Comparator Group
Number analyzed (Participants) | 70 | 70
participants | 12 | 6

ADVERSE EVENTS:
Time Frame: 2 year, 3 months. Adverse event tables presented include data reported through End Of Study
Description: An adverse event was defined as any noxious and unintended sign, symptom, or disease that began or worsened from the time the patient signed the Informed Consent Form to participate in the study until 30 days after last study treatment, regardless of whether event was considered related or unrelated to study drug. Treatment emergent adverse events were summarized in the table below (patients who received study drug - 68/67). NCI CTCAE V3 was used to assess toxicities observed during the study.
Arm/Group | Experimental Group | Comparator Group
All-Cause Mortality (participants affected / at risk) | 49/68 | 52/67
Serious Adverse Events (participants affected / at risk) | 35/68 | 30/67
Other Adverse Events (participants affected / at risk) | 66/68 | 61/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=68) | Comparator Group (N=67)
Neutropenia (Blood and lymphatic system disorders) | 9 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6
Anemia (Blood and lymphatic system disorders) | 2 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive Airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Venous Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 2
Circulatory Collapse (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 2 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 7
Asthenia (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Generalised Oedema (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Multi-organ Failure (General disorders) | 1 | 0
Non-cardiac Chest pain (General disorders) | 1 | 0
Performance Status Decreased (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 4
Cellulitis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 2 | 0
Candiddiasis (Infections and infestations) | 1 | 0
Catheter realted infection (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Gastroenteristic Salmonella (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Herpes Virus Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0
Blood Albumin Decreased (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 1 | 0
Urine Output Decreased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Abdominal Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1
Depressed level Of Consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 4
Obstructive Uropathy (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=68) | Comparator Group (N=67)
Anemia (Blood and lymphatic system disorders) | 21 | 22
Neutropenia (Blood and lymphatic system disorders) | 34 | 16
Leukopenia (Blood and lymphatic system disorders) | 17 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 13
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 5
Cardiac Disorders (Cardiac disorders) | 14 | 9 — Cardiac AEs are presented as a grouping within the SOC of Cardiac Disorders as no specific preferred term was reported > 5%. PTs include, but are not limited to, cardiac failure, left ventricular dysfunction and ejection fraction decreased.
Nausea (Gastrointestinal disorders) | 12 | 11
Abdominal Pain (Gastrointestinal disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 5 | 10
Diarrhea (Gastrointestinal disorders) | 3 | 12
Asthenia (General disorders) | 16 | 9
Pyrexia (General disorders) | 16 | 16
Edema peripheral (General disorders) | 10 | 4
Fatigue (General disorders) | 9 | 9
Mucosal inflammation (General disorders) | 8 | 2
Pneumonia (Infections and infestations) | 5 | 4
Bronchitis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 4 | 2
Ejection fraction decreased (Investigations) | 13 | 7
Weight Decreased (Investigations) | 5 | 5
Platelet count decreased (Investigations) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 8 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9
Chromaturia (Renal and urinary disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 3
Skin Discoloration (Skin and subcutaneous tissue disorders) | 7 | 0
Hypotension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less